CLINICAL TRIAL: NCT06267378
Title: Assessing Frailty and Its Impacts in Older Patients Facing Major Gastrointestinal Surgery
Brief Title: Assessing Frailty and Its Impacts on Patients Facing Major GI Surgery
Status: Recruiting | Type: Observational
Sponsor: Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1174/2022/NCTS
Record Dates: First submitted 2023-10-24; First posted 2024-02-20 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-10

CONDITIONS: Bowel Cancer
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and Tissue collection from the resected specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Frailty measure — All participants will be asked to complete baseline assessments and a blood test.
  30 participants out of the 100 will be selected to wear a digital motion device before their surgery for seven days. (15 participants will be non-frail and 15 patients will be frail).
  Where possible, all baseline assessments will be scheduled to coincide with a routine clinic/hospital visit. The first assessment will complete functional, frailty, nutritional, and quality of life questionnaires. A blood test will be taken for baseline tests and metabolomic assessment. Participants who opt into having a digital motion device will also be shown how to use the device and will wear this for seven days. Written instructions to fit the device will also be given.

SUMMARY:
The study team will look at 3 new tests that will make it easier to measure frailty in patients awaiting surgery for cancer and compare them against standard clinical measures of frailty in a pilot study. The expected outcome is that evidence will be collated in order to apply for a major grant to look at improving the care of frail patients with cancer in the future.

DETAILED DESCRIPTION:
Over 40% of patients with bowel cancer are over the age of 75. In older patients, rates of ill health and frailty are high, with frailty found in 6 in 10 patients over the age of 90. Surgery is the main treatment for bowel cancer, but the risks of surgery are higher in older people especially if they are frail. The main features of frailty are weight loss, lack of energy, weakness, slow walking speed and low activity levels. Frailty is a condition linked to an increased risk of death and major complications after surgery. As a result, older and frailer patients are often refused surgery for their cancer. If we could identify frailty more reliably before surgery, we could offer patients better counselling about the surgical risks and benefits. We could also offer treatments that might improve their fitness, making the surgery safer (pre-operative exercise, better post-operative support). Surgeons are not very good at measuring frailty because the clinical tests for it are complicated and take a long time to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Aged 70 years and over.
3. Patients with a diagnosis of primary operable colorectal cancer where treatment includes a planned curative surgical procedure.
4. About to undergo elective surgery for cancer.
5. Mental capacity to consent.

Exclusion Criteria:

1. Patients with unresectable cancer.
2. Patients presenting as an emergency.
3. Patients who are having chemotherapy or radiotherapy before their surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastrointestinal cancer patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The sensitivity & specificity of digital motion data for the prediction of baseline clinical frailty levels & post-operative measures of frailty, mortality and adverse events | 01/12/2029
  The development of biochemical assessments of frailty could also provide valuable information to guide the treatment of the older patient although there are very few that have been validated for clinical use across a range of settings.
The sensitivity & specificity of tissue senescence for the prediction of baseline clinical frailty levels & post-operative measures of frailty, mortality and adverse events | 01/12/2029
  A further potential measure of frailty is tissue levels of senescence. Senescent cells are rare in the tissues of young organisms but become more common as tissues age, especially in adipose tissue, muscle and skin (Tchkonia et al., 2010). Both ageing and frailty are associated with cellular senescence, a mechanism of irreversible cell cycle arrest caused by persistent stress and damage, which contributes to the process of ageing, frailty and a range of diseases (Xu et al., 2018; Hickson et al., 2019). Senescent cells are causal to a wide range of diseases such as arthritis, arteriosclerosis and dementia and are also linked to the development of frailty in animal models.
The sensitivity & specificity of blood based biomarkers for the prediction of baseline clinical frailty levels & post-operative measures of frailty, mortality and adverse events | 01/12/2029
  A simple, validated biomarker of frailty, capable of identification of patients who are at an increased risk of adverse outcomes from surgery, would be of great value in the surgical decision-making process.

SECONDARY OUTCOMES:
Blood biomarker correlation (baseline and post operative) with baseline frailty and poor outcomes (including length of stay and adverse events) | 01/12/2029
  as above
Adverse events related to surgery assessed CTCAE classifications | 01/12/2029
  as above
Tissue senescence correlation between baseline frailty and poor outcomes (including length of stay and adverse events) | 01/12/2029
  as above
Digital mobility outcomes correlation with baseline frailty and poor outcomes (including length of stay and adverse events) | 01/12/2029
  as above
Physical function assessment after surgery at 6 weeks, 3 months using the WHO DAS 2.0. | 01/12/2029
  as above
Quality of life at 6 weeks, 3 months after surgery using the EQ-5D-5L | 01/12/2029
  as above
Overall survival at 3 months and 5 years (the latter via cancer registry returns) | 01/12/2029
  as above

CONTACTS AND LOCATIONS:
Overall Officials: Jayan George, Principal Investigator — Doncaster & Bassetlaw Teaching Hospitals NHS Foundation Trust
Locations (1):
- Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
TBC